CLINICAL TRIAL: NCT02917226
Title: A Mobile and Web-Based Clinical Decision Support and Monitoring System for Diabetes Mellitus Patients in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Vildan Mevsim, Prof.Dr. Vildan MEVSİM, MD, PhD, Dokuz Eylul University
Other Study IDs: 2015/23-40
Record Dates: First submitted 2016-08-24; First posted 2016-09-28 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinical decision support and monitoring system (Experimental)
  Interventions: Other: Clinical decision support and monitoring system
- Control Group (No Intervention)

INTERVENTIONS:
Other: Clinical decision support and monitoring system
  Arms: Clinical decision support and monitoring system

SUMMARY:
The purpose of the study is to develop a user-friendly, comprehensive, fully integrated web and mobile-based Clinical Decision Support and Monitoring System (CDSMS) for DM diseases screening, diagnosis, treatment and monitoring for the use of physicians and patients in primary care and to determine the effectiveness of the system. For validating the CDSMS for diabetes patients, randomized controlled trial will be conducted.A parallel single blind randomized controlled trial will be implemented. 10 physicians and their 439 patients are involved in the study. According to the results of screening which is done using developed CDSMS, DM diagnosed patients will be recruited for trial from the primary care centers by the physicians. The recruited patients will register to the CDSMS with their accounts given by their physicians. Eligible participants will be assigned to intervention and control groups with simple randomization. The significance level will be accepted as p<0,05. In the intervention group, the system recommendations on diagnosis, treatment and monitoring will be carried out as the final decision given by the physician. In the control group, physicians will treat DM patients as the general routine. Patients in both groups will be monitored for 6 months. Patient data on 0th and 6th month will be compared. Clinical and laboratory outcomes will be face-to-face assessed, others will be online self-assessed.

ELIGIBILITY:
Inclusion Criteria:

* Being over age 40
* Volunteer
* Computer and Internet literacy
* DM diagnosed or having at least one of diagnostic criteria.

These criteria;

* HbA1c ≥ 6.5
* FPG ≥ 126 mg / dl
* 2-hour postprandial glucose ≥ 200 mg / dl
* Any time postprandial glucose ≥ 200 mg / dl
* Diabetes symptoms

Exclusion Criteria:

* Having a communication problem
* Type 1 diabetes
* MODY type DM
* Level of psychiatric disorders in psychosis
* Dementia ones

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
fasting blood glucose | Change from baseline fasting blood glucose at 6 months

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kart O, Mevsim V, Kut A, Yurek I, Altin AO, Yilmaz O. A mobile and web-based clinical decision support and monitoring system for diabetes mellitus patients in primary care: a study protocol for a randomized controlled trial. BMC Med Inform Decis Mak. 2017 Nov 29;17(1):154. doi: 10.1186/s12911-017-0558-6. PMID 29187186